CLINICAL TRIAL: NCT02289612
Title: The Pudding Study: The Effect of Effect of Fibre-enriched Pudding Products on Glycemic and Satiety Response in Adults at Risk for Type 2 Diabetes
Brief Title: Glycemic and Satiety Response Study of Fibre-Enriched Pudding Products
Acronym: Pudding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Ontario Ministry of Agriculture, Food and Rural Affairs (Other Government); Natural Sciences and Engineering Research Council, Canada (Other); Dairy Farmers of Ontario (Other); Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Principal Investigator, Alison Duncan, Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 14AP003; 200603 (Other Grant/Funding Number: OMAFRA)
Record Dates: First submitted 2014-11-05; First posted 2014-11-13 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Risk for Type 2 Diabetes Mellitus; Fibre; Postprandial Glucose; Postprandial Insulin; Postprandial Acetaminophen; Satiety
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Tapioca Starch - Low-Fibre (Placebo Comparator): Tapoica starch pudding without added fibre
  Interventions: Other: Yellow Mustard Gum Fibre
- High Maltose Corn Syrup - Low-Fibre (Placebo Comparator): High maltose corn syrup pudding without added fibre
  Interventions: Other: Yellow Mustard Gum Fibre
- Trutol Glucose Beverage (#1) (Placebo Comparator): Trutol Glucose Beverage containing 50 g of glucose without added fibre. Consumed at first treatment study visit.
  Interventions: Other: Yellow Mustard Gum Fibre
- Trutol Glucose Beverage (#2) (Placebo Comparator): Trutol Glucose Beverage containing 50 g of glucose without added fibre. Consumed at final treatment study visit.
  Interventions: Other: Yellow Mustard Gum Fibre
- Yellow Mustard Gum Fibre - Tapioca Starch (Active Comparator): Yellow mustard gum fibre pudding containing tapioca starch. Fibre-enriched treatment product.
  Interventions: Other: Yellow Mustard Gum Fibre
- Yellow Mustard Gum Fibre - High Maltose Corn Syrup (Active Comparator): Yellow mustard gum fibre pudding containing high maltose corn syrup. Fibre-enriched treatment product.
  Interventions: Other: Yellow Mustard Gum Fibre
- Soluble Flaxseed Gum Fibre - Tapioca Starch (Active Comparator): Soluble flaxseed gum fibre pudding containing tapioca starch. Fibre-enriched treatment product.
  Interventions: Other: Soluble Flaxseed Gum Fibre
- Soluble Flaxseed Gum Fibre - High Maltose Corn Syrup (Active Comparator): Soluble flaxseed gum fibre pudding containing high maltose corn syrup. Fibre-enriched treatment product.
  Interventions: Other: Soluble Flaxseed Gum Fibre
- Fenugreek Gum Fibre - Tapioca Starch (Active Comparator): Fenugreek gum fibre pudding containing tapioca starch. Fibre-enriched treatment product.
  Interventions: Other: Fenugreek Gum Fibre
- Fenugreek Gum Fibre - High Maltose Corn Syrup (Active Comparator): Fenugreek gum fibre pudding containing high maltose corn syrup. Fibre-enriched treatment product.
  Interventions: Other: Fenugreek Gum Fibre

INTERVENTIONS:
Other: Yellow Mustard Gum Fibre
  Arms: High Maltose Corn Syrup - Low-Fibre; Tapioca Starch - Low-Fibre; Trutol Glucose Beverage (#1); Trutol Glucose Beverage (#2); Yellow Mustard Gum Fibre - High Maltose Corn Syrup; Yellow Mustard Gum Fibre - Tapioca Starch
Other: Soluble Flaxseed Gum Fibre
  Arms: Soluble Flaxseed Gum Fibre - High Maltose Corn Syrup; Soluble Flaxseed Gum Fibre - Tapioca Starch
Other: Fenugreek Gum Fibre
  Arms: Fenugreek Gum Fibre - High Maltose Corn Syrup; Fenugreek Gum Fibre - Tapioca Starch

SUMMARY:
The purpose of this study is to determine the specific properties of a variety of dietary fibres that lead to different postprandial glycemic and satiety responses in individuals at risk for type 2 diabetes. This is accomplished by utilizing a variety of dietary fibres that demonstrate a wide range of properties in a pudding product, and by examining the ability of each of these to limit gastric emptying, limit glucose absorption, limit insulin secretion, and improve satiety, versus a low fibre control product.

DETAILED DESCRIPTION:
The purpose of this study is to determine the specific properties of a variety of dietary fibres that lead to different postprandial glycemic and satiety responses in individuals at risk for type 2 diabetes. This is accomplished by utilizing a variety of dietary fibres that demonstrate a wide range of properties in a pudding product, and by examining the ability of each of these to limit gastric emptying, limit glucose absorption, limit insulin secretion, and improve satiety, versus a low fibre control product. To accomplish this, a randomized, double-blinded, placebo controlled, crossover study design will be used, in order to determine the different effects of a variety of fibre-enriched pudding products on markers of type 2 diabetes and satiety response, versus low-fibre control puddings.

ELIGIBILITY:
Inclusion Criteria:

* Men/Women
* Age 18-70 years
* CANRISK Questionnaire score ≥21 (brief questionnaire that identifies risk of diabetes)
* BMI ≥25 and <40 kg/m2
* Prior use of acetaminophen

Exclusion Criteria:

* Smokers
* Food allergies or any life-threatening allergy (food or otherwise)
* Acetaminophen allergy
* Gastrointestinal conditions or illnesses (Including, but not limited to, lactose intolerance, Celiac, Crohn's, Ulcerative Colitis (UC), Irritable Bowel Disorder (IBD))
* Serious major medical condition (i.e. renal, liver)
* Pregnant or breastfeeding
* Food Neophobia Scale score between 30 and 54 (Food Neophobia Scale is a questionnaire which is intended to screen out individuals who are unsure of consuming new products)
* TFEQ-CR >16 (TFEQ is a questionnaire to screen for restrained eaters)
* Alcohol consumption>4 drinks/sitting
* Medication or natural health products (NHPs) used for diabetes (glycemic control)
* Medication or NHPs contraindicated with acetaminophen
* Recent or intended significant weight loss or gain (i.e. >4 kg in previous 3 months)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Fasting and postprandial blood glucose response for each pudding and control product | Blood glucose will be analyzed for each study visit (10 in total) at times 0 (fasting), 15, 30, 60, 90, and 120 minutes, to compare responses between different treatment products.
  Blood glucose will be measured in the fasting state and postprandially through finger prick blood samples at each study visit. Participants will have an initial fasted blood sample taken, then consume one of 10 treatment products over a 10 minute period, and will then have blood taken at 15, 30, 60, 90, and 120 minute intervals. This will occur once a week for 10 weeks until all treatments have been consumed.
Fasting and postprandial insulin response for each pudding and control product | Blood insulin will be analyzed for each each study visit (10 in total), at times 0 (fasting), 15, 30, 60, 90, and 120 minutes, to compare responses between different treatment products.
  Insulin will be measured in the fasting state and postprandially through finger prick blood samples at each study treatment visit. Participants will have an initial fasted blood sample taken, then consume one of 10 treatment products over a 10 minute period, and will then have blood taken at 15, 30, 60, 90, and 120 minute intervals. This will occur once a week for 10 weeks until all treatments have been consumed.
Fasting and postprandial acetaminophen absorption for each pudding and control product | Blood acetaminophen will be analyzed for each study visit (10 in total) at times 0 (fasting), 15, 30, 60, 90, and 120 minutes, to compare responses between different treatment products.
  Acetaminophen will be measured in the fasting state and postprandially through finger prick blood samples at each study treatment visit. Participants will have an initial fasted blood sample taken, then consume one of 10 treatment products over a 10 minute period, and will then have blood taken at 15, 30, 60, 90, and 120 minute intervals. This will occur once a week for 10 weeks until all treatments have been consumed.
Satiety-producing effect for each pudding and control product | Satiety will be analyzed for each study visit (10 in total) at times 0 (fasting), 15, 30, 60, 90, and 120 minutes, to compare responses between different treatment products.
  Participants will complete visual analogue scale (VAS) questionnaires during each treatment visit to subjectively measure satiety. They will be asked to complete an initial VAS questionnaire when fasted, and will then consume one of 10 treatments within 10 minutes, and complete VAS questionnaires 5 minutes before each blood sample at times 10, 25, 55, 85, and 115 minutes. After 120 minutes have passed, participants will consume an ad libitum pizza lunch buffet meal to objectively measure satiety, and once comfortably full they will complete a final VAS questionnaire. Weighed food records will be used to objectively measure food intake for the rest of the day. This will occur once a week for 10 weeks until all treatments have been consumed.

SECONDARY OUTCOMES:
3-Day food records | Over 3 days before the first treatment study visit
  Participants will complete 3-day food records before the first treatment study visit to provide information about their background nutrient intake and dietary habits.

OTHER OUTCOMES:
Fasted body weight | At each study treatment visit
  Fasted body weight will be measured at each study before consuming the treatment product.
Heart rate and blood pressure | At each study treatment visit
  Heart rate (beats per minute) and blood pressure (systolic/diastolic mmHg) will be measured at each study treatment visit before consuming the treatment product.

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Duncan, Ph.D., R.D., Principal Investigator — University of Guelph, Human Nutraceutical Research Unit; Amanda J Wright, Ph.D., Study Director — University of Guelph, Human Nutraceutical Research Unit; Alison M Duncan, Ph.D., R.D., Study Director — University of Guelph, Human Nutraceutical Research Unit
Locations (1):
- Human Nutraceutical Research Unit, Guelph, Ontario, Canada